CLINICAL TRIAL: NCT04861558
Title: EFFIPEC - Efficacy of Hyperthermic Intraperitoneal Chemotherapy, Single-arm Phase I Study, Followed by an Open-label, Randomized, Controlled Registry-based Phase III Trial
Brief Title: Efficacy of Hyperthermic Intraperitoneal Chemotherapy
Acronym: EFFIPEC
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Uppsala University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: EFFIPECv5
Record Dates: First submitted 2021-04-06; First posted 2021-04-27 (Actual); Last update posted 2025-05-30 (Actual); Status verified 2025-05

CONDITIONS: Colorectal Cancer; Peritoneal Metastases
MeSH Terms: conditions — Colorectal Neoplasms | interventions — Fluorouracil; Irinotecan; Oxaliplatin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Standard HIPEC (Active Comparator): Injection of oxaliplatin 460 mg/m2 and an intraoperational IV of 5-fluorouracil 400 mg/m2, and calcium folinate 60 mg/m2.
  Interventions: Drug: Oxaliplatin
- Intensified HIPEC+EPIC (Experimental): Injection of irinotecan 360 mg/m2 and 5-fluorouracil 24-hr EPIC 250-850 mg/m2 in combination with Oxaliplatin 360 mg/m2 and an intraoperational IV of 5-fluorouracil bolus 400 mg/m2 with calcium folinate 60mg/m2.
  The EPIC treatment is given after the abdomen is completely sutured in the operating theater. The dose will be divided equally into 2 injections á 200ml each through two abdominal drains.
  Interventions: Drug: 5Fluorouracil; Drug: Irinotecan; Drug: Oxaliplatin

INTERVENTIONS:
Drug: 5Fluorouracil — Injection of 250-850 mg/m2.
  Other Names: Fluorouracil Accord; Fluorouracil Tevo
  Arms: Intensified HIPEC+EPIC
Drug: Irinotecan — Injection of 360 mg/m2
  Other Names: Irinotecan Accord; Irinotecan Actavis; Irinotecan Fresenius Kabi
  Arms: Intensified HIPEC+EPIC
Drug: Oxaliplatin — Injection of 460 mg/m2
  Other Names: Oxaliplatin Accord; Oxaliplatin Teva; Oxaliplatin Fresenius Kabi

SUMMARY:
A dose titration study and a combined superiority registry-based open-label randomized control trial is planned to answer the trial objectives. The study will be registry-based to allow simpler and more comprehensive follow-up. Patients with colorectal cancer will be treated with cytoreductive surgery (CRS) together with either standard oxaliplatin HIPEC (the control for the efficacy study) or oxaliplatin/irinotecan HIPEC in combination with 5-FU 24-hour EPIC. The 5-FU will be administered postoperatively when the abdomen is completely sutured. The drug is divided equally into 2 injections of 200 ml each and injected through two abdominal drains that are clamped for 16 hours.

For dose escalation, the titration groups (á 3 or 6 patients) are followed for 30 days postoperatively after which the Data Monitoring Committee (DMC) will determine whether or not to increase the 5-FU dose for the following group of patients.

To study efficacy, randomization is performed intraoperatively. The patient is followed up postoperatively for a total of 3 years for the secondary endpoints which may be extended by the study committee to 5 years. Since the trial is registry based, the long-term follow-up does not require separate eCRF evaluations. These evaluations can be automatically retrieved from the registry - both recurrence data, quality of life, and morbidity data. Some specific eCRF evaluations will be integrated as a separate study part of the HIPEC registry, such as inclusion/exclusion criteria and adverse event reporting (including SUSAR reporting).

DETAILED DESCRIPTION:
Not detailed description entered.

ELIGIBILITY:
Inclusion criteria:

1. Provision of written informed consent prior to any study specific procedures.
2. ECOG Performance Status Score 0,1 or 2 alternatively Karnofsky 60-100
3. Adequate kidney, liver, bone marrow function according to laboratory tests
4. For females of childbearing potential, a negative pregnancy test must be documented
5. ≥ 18 years old and ≤78 years old
6. Colorectal cancer with peritoneal metastases +/- liver metastases (maximum 3)
7. Concomitant resectable pulmonary metastases are allowed
8. All patients deemed eligible for CRS and HIPEC according to clinical routine management during a HIPEC multidisciplinary board at each respective hospital can be included.

Exclusion criteria:

1. Previous severe toxicity/allergic reactions to systemic chemotherapy agents oxaliplatin or irinotecan or 5-fluorouracil
2. Unable to tolerate intensified HIPEC treatment due to comorbidity
3. Metastasis other than peritoneum or liver or lung
4. Complex liver-perenchymal sparing surgery or hemihepatectomy procedures are to be excluded.
5. Previous CRS or HIPEC
6. Pregnant or lactating (nursing) women
7. Active infections requiring antibiotics
8. Active liver disease with positive serology for active hepatitis B, C, or known HIV
9. Concurrent administration of any cancer therapy other than planned study treatment within 4 weeks prior to and up to 4 weeks after study treatment
10. Incomplete cytoreduction defined as completeness of cytoreduction score 2-3
11. Histopathology of other origin than colorectal cancer

Ages: 18 Years to 79 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 213 (Estimated)
Dates: Start 2021-05-01 (Actual); Primary Completion 2025-12 (Estimated); Study Completion 2029-12 (Estimated)

PRIMARY OUTCOMES:
Recurrence-free survival | 24 months after treatment
  To study the recurrence-free survival (RFS) of patients

SECONDARY OUTCOMES:
Overall survival | 5 years after treatment
  Survival is followed through the HIPEC registry.
Recurrence-free survival | 5 years after treatment
  Survival is followed through the HIPEC registry. The RECIST criteria are used to determine recurrence and site of first recurrence
Postoperative complication rate | Within 30 days after treatment
  Morbidity is registered in the HIPEC registry within 30 days of treatment administration.
Patient evaluations of quality of life | 3 years after treatment
  EORTC QLQ questionnaire filled out at baseline, 12 and 36 months after surgery using the established QoL database.

CONTACTS AND LOCATIONS:
Overall Officials: Peter Cashin, MD, PhD, Principal Investigator — Uppsala University Hospital
Locations (5):
- INDEPSO, Ahmedabad, India
- Sweden (4):
  - Sahlgrenska östra sjukhuset, Gothenburg
  - Skånes universitetssjukhus, Malmo
  - Karolinska sjukhuset, Stockholm
  - Akademiska sjukhuset, Uppsala

IPD SHARING:
Plan to Share IPD: Yes
Completely anonymized IPD will be shared. All dates, HIPEC center treatment, referral city, and personal identification will be removed.
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: To be shared at the time of phase 3 trial publication. Available for 10 years.
Access Criteria: Access by request only from the corresponding author. Study protocol, SAP, ICF will be publicly available without request.